CLINICAL TRIAL: NCT04855578
Title: GABA-WHY Study: Deprescription of Gabapentinoids in Medical Inpatients
Brief Title: Deprescription of Gabapentinoids in Medical Inpatients
Acronym: GABA-WHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Dr. Emily McDonald, Associate Professor of Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-7353
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Polypharmacy; Gabapentin; Pregabalin
Keywords: Polypharmacy; Deprescribing; Gabapentin; Pregabalin; Medication Stewardship; High-Value Healthcare; Empowerment; Shared Decision-Making; Adverse Drug Reaction; Elderly; Frailty
MeSH Terms: conditions — Empowerment; Drug-Related Side Effects and Adverse Reactions; Frailty

STUDY DESIGN:
Intervention Model Description: Prospective before-and-after study involving five medical wards at two health centres. All wards will start in the control phase and enrolled participants will receive standard therapy. Once the pre-specified target of a 80 participants have been enrolled, all five wards will simultaneously transition into the intervention phase. All subsequently enrolled participants will receive the intervention until another 80 participants are enrolled. The control and intervention phases are expected to take approximately 5 months each.
Who Masked: Investigator
Masking Description: It is impossible to blind physicians or study participants. However, medical staff on study units will not be told that gabapentinoids are being targeted by the trial until after the control period has ended. The rationale is that prior knowledge of the goal may bias medical staff in favour of gabapentinoid deprescription. Similarly, participants recruited during the control period will not be told that gabapentinoids are targeted. Since medical staff work in multiple study units in a given year, all units will transition from the control phase to the intervention phase simultaneously to prevent contamination between the control and intervention group.
  It is impossible to blind outcome assessors at the time of follow-up. Undue influence on the investigator by outcome assessors will be mitigated through the use of a standardized survey that do not depend on the judgement of outcome assessors. Additionally, patient data will be anonymized with a unique identifier prior to analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Medical Care (No Intervention): During the control period, patients admitted to the study sites who qualify for the trial will receive a pharmacy medication reconciliation as part of usual medical care. Study participants will be informed that the goal of the trial is to evaluate medication use and medication changes after discharge, but they will not be informed that gabapentinoids are specifically being targeted. Medical staff will not receive specific information about the trial, or particular instructions with regards to deprescription during the control period.
- In-Hopsital Patient Educational Brochure and Physician Education about Gabapentinoid Prescription (Experimental): During the intervention period, patients admitted to the study sites who qualify for the trial will receive an in-hospital educational brochure. Additionally, the medical team will attend an educational session about gabapentinoid prescription.
  Interventions: Other: In-Hopsital Patient Educational Brochure; Other: Physician Education about Gabapentinoid Prescription

INTERVENTIONS:
Other: In-Hopsital Patient Educational Brochure — The participant's medication list will be identified from the pharmacy database and validated with the participant's best possible medication history taken at time of admission by a pharmacist. Eligibility will be confirmed by the participant's treating medical team with support from the study investigators. Participants who are enrolled during the intervention phase will receive an educational brochure about the risks of chronic gabapentinoid use, and about how to safely discontinue use. The brochure is written using a sixth-grade vocabulary and has been validated in both English and French for comprehension and readability, including for people with mild cognitive impairment.
  Arms: In-Hopsital Patient Educational Brochure and Physician Education about Gabapentinoid Prescription
Other: Physician Education about Gabapentinoid Prescription — An educational session about the purpose of the study and risks of gabapentinoid prescription will be delivered to physicians (staff and medical residents) on each study unit at both sites during the intervention period. The educational session will include a presentation by the chief of the medical service at the monthly teaching rounds, and an electronic message will be sent to all physicians on the medical service. Physicians will also be presented a brief overview of the educational brochure.
  Arms: In-Hopsital Patient Educational Brochure and Physician Education about Gabapentinoid Prescription

SUMMARY:
In this trial, investigators will distribute educational brochures with information about the deprescription of gabapentinoids (gabapentin and pregabalin) to inpatients in five medical wards spread across two tertiary-care hospitals in Montréal, Canada. This intervention will be supplemented by a brief information session for medical staff on the wards. This study aims to evaluate the effectiveness of this combined intervention on increasing gabapentinoid deprescription rates among study participants compared to control following hospital discharge.

DETAILED DESCRIPTION:
Gabapentinoids, which include gabapentin and pregabalin, are antiepileptic drugs that have been approved by the FDA and Health Canada for the treatment of postherpetic neuralgia, with pregabalin also approved for the treatment of diabetic neuropathy, fibromyalgia, and spinal cord injury-associated neuropathic pain. Despite a small number of approved indications, gabapentinoid prescription has increased substantially in recent years. The majority of new prescriptions are off-label for the treatment of multiple chronic pain conditions, such as osteoarthritis, chronic lower back pain, sciatica, and cancer-related pain.

A 2013 Cochrane review found reasonably good evidence for the use of both drugs in postherpetic neuralgia and painful diabetic neuropathy, as well as evidence supporting pregabalin use for the treatment of fibromyalgia and central neuropathic pain. However, there was either evidence against, or a lack of evidence for the efficacy of gabapentinoids in other chronic pain conditions. Furthermore, beneficial effects were associated with high risk of multiple adverse effects, including sedation, xerostomia, lower extremity edema, and traumatic falls in older adults.

In a recent study of inpatients at a tertiary-care hospital in Montréal, Canada between 2013 and 2017, 1 in 8 patients had a gabapentinoid prescription on admission, only 17% of which were for an FDA-approved indications. Gabapentinoid users had more comorbidities than non-users and were more likely to be co-prescribed opioids, which is concerning given previous evidence of increased opioid-related death with gabapentinoid co-prescriptions. Given their high prevalence of off-label use, their many adverse effects, and their frequent use among multimorbid patients who are vulnerable to these adverse effects, gabapentinoids are an ideal target for deprescription.

Patient education through the distribution of educational brochures is an effective method of promoting deprescription. A brochure specific to gabapentinoids is available on the Canadian Deprescribing Network website. This brochure contains a self-assessment of knowledge of the risks of gabapentinoids, provides information on the benefits and potential harms of use, presents safer treatment alternatives, and proposes a tapering regimen using an illustrated calendar, with instructions to contact a healthcare provider prior to discontinuation or tapering. This brochure aims to improve safe and successful deprescription by promoting patient motivation and self-capacity, and by encouraging patients to meet with their healthcare providers to create opportunities for deprescription.

In previous studies, a similar brochure was found effective in promoting benzodiazepine deprescription. In the Eliminating Medications through Patient Ownership of End Results (EMPOWER) trial, the distribution of educational brochures to 303 community-dwelling older adults who were chronically taking benzodiazepines resulted in a 27% discontinuation rate at 6 months, compared to a 5% discontinuation rate in the control group. The EMPOWER trial inspired a subsequent study in which the same brochure was distributed to medical inpatients at a tertiary-care hospital in Montreal, Canada. A total of 50 patients received the brochure while hospitalized, and 64% of those patients had discontinued benzodiazepines at 30 days-post discharge. This result was significantly higher than the hospital's historical deprescription rate of 21%. The higher deprescription rate associated with the intervention in this study compared to the EMPOWER trial highlights the importance of using hospital admissions as an opportunity for deprescription. Thus, the aim of this trial is to assess the efficacy of an educational brochure about gabapentinoids in improving gabapentinoid deprescription among elderly inpatients after discharge.

This study will follow a prospective controlled before and after study design involving five medical units across two centres: the McGill University Health Centre Glen Site (Royal Victoria Hospital) and the Montreal General Hospital. The sample size of the study is 160 participants, with 80 participants in the control group and 80 participants in the intervention group. The sample size was calculated to detect a 20% absolute increase in deprescription within the intervention group. Each study unit will act as its own control. The study will begin in the control period on all study units, until the pre-specified target of 80 control participants are enrolled. Once the enrolment of the 80 control participants has been completed, all study units will simultaneously transition to the intervention period. The intervention period will be completed once the pre-specified target number of 80 intervention participants is reached. Recruitment is expected to last approximately 10 months, with 16 patients enrolled per month. This rate of enrolment is based on previous study data regarding the prevalence of admitted gabapentinoid users and historical admission statistics from the study units, and assumes a study participation refusal rate of 15%.

During the control period, enrolled patients admitted to the medical ward will receive a pharmacy medication reconciliation as part of usual medical care. Although they will be informed that the goal of the trial is to evaluate medications and changes after discharge, participants will not be told that gabapentinoids are specifically being targeted. Additionally, medical staff will not receive specific information about the trial, or particular instructions related to deprescription.

During the intervention period, enrolled patients will receive an educational brochure about the risks of chronic gabapentinoid use and how to safely discontinue use. The educational brochure is written using a sixth-grade vocabulary and has been validated in both English and French for comprehension among individuals with and without mild cognitive impairment. Additionally, an educational session detailing purpose of the study and the risks of gabapentinoid prescription will be delivered to medical staff and residents on each study unit. The educational session will include a presentation by the chief of the medical service at the monthly teaching rounds, and an electronic message sent to all physicians on the medical service. The session will also include a brief overview of the brochure.

Follow-up questionnaires will be administered at 8 weeks after hospital discharge by telephone. The questionnaire will collect information regarding demographic changes, gabapentinoid deprescription, use of other pain medications, withdrawal symptoms, global functioning, pain control, and cognition.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients 60 years or older admitted to study units who have a gabapentinoid prescription prior to admission

Exclusion Criteria:

* Less than 60 years of age
* Known seizure disorder
* Not enrolled in the provincial drug plan (RAMQ)
* Opting out of the provincial drug database (Dossier Santé Québec), which will be confirmed with the patient at the time of recruitment
* Previous enrollment in the study
* Patients expected to die before primary endpoint can be realized (e.g., patients admitted for end-of-life care or prognosis of 3 months or less)
* Unable to consent
* Major neurocognitive disorder, as determined by a previously established diagnosis or interim diagnosis by the medical staff on the ward of moderate severity or worse
* Unable to speak English or French
* Insufficient literacy in English or French
* No means of contacting patient by phone after discharge (e.g. no valid phone number, traveling, planned discharge to a facility without means of reaching by phone, etc.)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Gabapentinoid Discontinuation or Dose Reduction With Intention to Stop | 8-weeks post-hospital discharge
  Proportion of study participants with a gabapentinoid prescription stopped or decreased with intention to stop at the time of follow-up

SECONDARY OUTCOMES:
Gabapentinoid Dose Reduction Without Intention to Stop | 8-weeks post-hospital discharge
  Proportion of study participants with a gabapentinoid dose reduction without intention to stop at the time of follow-up
Health and Global Function | At study enrollment and 8-weeks post-hospital discharge
  Assessed by the Patient Reported Outcomes Measurement and Information System (PROMIS) scale v1.2 - Global Health. This scale consists of four questions that are scored from 1 to 5, where higher scores indicate better health and global function.
Chronic Pain Intensity | At study enrollment and 8-weeks post-hospital discharge
  Assessed by the Patient Reported Outcomes Measurement and Information System (PROMIS) scale v2.0 - Pain Intensity 3a. This scale consists of three questions that are scored from 1 to 5, where higher scores indicate higher pain intensity.
Cognition | At study enrollment and 8-weeks post-hospital discharge
  Assessed by the Patient Reported Outcomes Measurement and Information System (PROMIS) scale v2.0 - Cognitive Function - Short Form 6a. This scale consists of six questions that are scored from 1 to 5, where higher scores indicate worse cognition.
Initiation of New Pain Medication | 8-weeks post-hospital discharge
  Proportion of study participants prescribed a new pain medication at the time of follow-up
Increase in Doses of Current Pain Medication | 8-weeks post-hospital discharge
  Proportion of study participants with an increase in dose of a non-gabapentinoid pain medication at the time of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Emily G McDonald, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Montreal General Hospital, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available in an anonymized format by emailing the primary investigator
Time Frame: One year following the primary publication
Access Criteria: Non-industry researchers

REFERENCES:
- [Background] Wilson MG, Lee TC, Hass A, Tannenbaum C, McDonald EG. EMPOWERing Hospitalized Older Adults to Deprescribe Sedative Hypnotics: A Pilot Study. J Am Geriatr Soc. 2018 Jul;66(6):1186-1189. doi: 10.1111/jgs.15300. Epub 2018 Mar 1. PMID 29492957
- [Background] Bennett MI, Laird B, van Litsenburg C, Nimour M. Pregabalin for the management of neuropathic pain in adults with cancer: a systematic review of the literature. Pain Med. 2013 Nov;14(11):1681-8. doi: 10.1111/pme.12212. Epub 2013 Aug 5. PMID 23915361
- [Background] Mathieson S, Maher CG, McLachlan AJ, Latimer J, Koes BW, Hancock MJ, Harris I, Day RO, Billot L, Pik J, Jan S, Lin CC. Trial of Pregabalin for Acute and Chronic Sciatica. N Engl J Med. 2017 Mar 23;376(12):1111-1120. doi: 10.1056/NEJMoa1614292. PMID 28328324
- [Background] Moore A, Derry S, Wiffen P. Gabapentin for Chronic Neuropathic Pain. JAMA. 2018 Feb 27;319(8):818-819. doi: 10.1001/jama.2017.21547. PMID 29486015
- [Background] Shanthanna H, Gilron I, Rajarathinam M, AlAmri R, Kamath S, Thabane L, Devereaux PJ, Bhandari M. Benefits and safety of gabapentinoids in chronic low back pain: A systematic review and meta-analysis of randomized controlled trials. PLoS Med. 2017 Aug 15;14(8):e1002369. doi: 10.1371/journal.pmed.1002369. eCollection 2017 Aug. PMID 28809936
- [Background] Wiffen PJ, Derry S, Bell RF, Rice AS, Tolle TR, Phillips T, Moore RA. Gabapentin for chronic neuropathic pain in adults. Cochrane Database Syst Rev. 2017 Jun 9;6(6):CD007938. doi: 10.1002/14651858.CD007938.pub4. PMID 28597471
- [Background] Wiffen PJ, Derry S, Moore RA, Aldington D, Cole P, Rice AS, Lunn MP, Hamunen K, Haanpaa M, Kalso EA. Antiepileptic drugs for neuropathic pain and fibromyalgia - an overview of Cochrane reviews. Cochrane Database Syst Rev. 2013 Nov 11;2013(11):CD010567. doi: 10.1002/14651858.CD010567.pub2. PMID 24217986
- [Background] Jette N, Lix LM, Metge CJ, Prior HJ, McChesney J, Leslie WD. Association of antiepileptic drugs with nontraumatic fractures: a population-based analysis. Arch Neurol. 2011 Jan;68(1):107-12. doi: 10.1001/archneurol.2010.341. PMID 21220681
- [Background] Toth C. Drug safety evaluation of pregabalin. Expert Opin Drug Saf. 2012 May;11(3):487-502. doi: 10.1517/14740338.2012.677026. Epub 2012 Apr 3. PMID 22468635
- [Background] Johansen ME. Gabapentinoid Use in the United States 2002 Through 2015. JAMA Intern Med. 2018 Feb 1;178(2):292-294. doi: 10.1001/jamainternmed.2017.7856. PMID 29297045
- [Background] Kwok H, Khuu W, Fernandes K, Martins D, Tadrous M, Singh S, Juurlink DN, Gomes T. Impact of Unrestricted Access to Pregabalin on the Use of Opioids and Other CNS-Active Medications: A Cross-Sectional Time Series Analysis. Pain Med. 2017 Jun 1;18(6):1019-1026. doi: 10.1093/pm/pnw351. PMID 28340102
- [Background] Hamer AM, Haxby DG, McFarland BH, Ketchum K. Gabapentin use in a managed medicaid population. J Manag Care Pharm. 2002 Jul-Aug;8(4):266-71. doi: 10.18553/jmcp.2002.8.4.266. PMID 14613419
- [Background] Scott IA, Hilmer SN, Reeve E, Potter K, Le Couteur D, Rigby D, Gnjidic D, Del Mar CB, Roughead EE, Page A, Jansen J, Martin JH. Reducing inappropriate polypharmacy: the process of deprescribing. JAMA Intern Med. 2015 May;175(5):827-34. doi: 10.1001/jamainternmed.2015.0324. PMID 25798731
- [Background] Martin P, Tannenbaum C. A realist evaluation of patients' decisions to deprescribe in the EMPOWER trial. BMJ Open. 2017 May 4;7(4):e015959. doi: 10.1136/bmjopen-2017-015959. PMID 28473524
- [Background] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Background] Martin P, Tannenbaum C. Use of the EMPOWER brochure to deprescribe sedative-hypnotic drugs in older adults with mild cognitive impairment. BMC Geriatr. 2017 Jan 31;17(1):37. doi: 10.1186/s12877-017-0432-5. PMID 28143413
- [Background] McDonald EG, Wu PE, Rashidi B, Forster AJ, Huang A, Pilote L, Papillon-Ferland L, Bonnici A, Tamblyn R, Whitty R, Porter S, Battu K, Downar J, Lee TC. The MedSafer Study: A Controlled Trial of an Electronic Decision Support Tool for Deprescribing in Acute Care. J Am Geriatr Soc. 2019 Sep;67(9):1843-1850. doi: 10.1111/jgs.16040. Epub 2019 Jun 27. PMID 31250427
- [Background] Gingras MA, Lieu A, Papillon-Ferland L, Lee TC, McDonald EG. Retrospective Cohort Study of the Prevalence of Off-label Gabapentinoid Prescriptions in Hospitalized Medical Patients. J Hosp Med. 2019 Sep;14(9):547-550. doi: 10.12788/jhm.3203. PMID 31112498
- [Derived] Williams J, Gingras MA, Dube R, Lee TC, McDonald EG. Patient empowerment brochures to increase gabapentinoid deprescribing: protocol for the prospective, controlled before-and-after GABA-WHY trial. CMAJ Open. 2022 Jul 12;10(3):E652-E656. doi: 10.9778/cmajo.20210302. Print 2022 Jul-Sep. PMID 35820684
- See also: Lyrica - Highlights of prescribing Information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2012/021446s028lbl.pdf
- See also: Neurontin - Highlights of prescribing Information — https://www.accessdata.fda.gov/drugsatfda_docs/label/2017/020235s064_020882s047_021129s046lbl.pdf
- See also: Lyrica - Product Monograph — https://pdf.hres.ca/dpd_pm/00070660.PDF
- See also: Neurontin - Product Monograph — https://pdf.hres.ca/dpd_pm/00044022.PDF
- See also: Canadian Deprescribing Network Patient Education Brochure - Gabapentinoids — https://static1.squarespace.com/static/5836f01fe6f2e1fa62c11f08/t/5f4f9501ca1e2c27719f7a77/1599051021132/Gabapentinoids_EN_Brochure.pdf